CLINICAL TRIAL: NCT02041143
Title: Effects of Protein Intake on Muscle Protein Synthesis and Whole Body Protein Balance During an Overnight Fast: an Exploratory Study
Brief Title: Protein Intake on Muscle Protein Synthesis Overnight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 13.19.MET
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Protein Synthesis Overnight
MeSH Terms: interventions — Milk Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milk protein (Experimental): Study product will provide 25 g of protein to subjects. One single supplement will be taken.
  Interventions: Dietary Supplement: Placebo
- Placebo (Placebo Comparator): Placebo (no protein)
  Interventions: Dietary Supplement: Milk protein

INTERVENTIONS:
Dietary Supplement: Milk protein — Study product will provide 25 g of protein to subjects.
  Arms: Placebo
Dietary Supplement: Placebo — Product with no protein
  Arms: Milk protein

SUMMARY:
This trial is an exploratory study in order to determine whether the ingestion of one type of protein (milk protein/CHO/Fat) vs.placebo (CHO/Fat) 2 hours before bed time results in the extension of the post-prandial window of anabolism during the night by increasing whole body protein balance as well as muscle protein fractional synthesis rate (FSR).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy as determined by the medical questionnaire and the medical visit including blood sampling
* 55-65y of age
* BMI (19.0 - 25.0 kg/ m²)
* Having signed the consent form

Exclusion Criteria:

* Digestive (intestinal, gastric, hepatic or pancreatic), renal or metabolic disease, as determined by the medical (screening) visit and a blood chemistry analysis (glucose, total cholesterol, LDL, HDL, triglycerides, aspartate transaminase, alanine aminotransferase, gamma glutamyl transpeptidase, C Reactive Protein, creatinin)
* Heart or other organ disease
* Arterial hypertension (Systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg)
* Any clotting trouble (diagnosed by Prothrombin time (PT), activated Partial Thromboplastin Time (aPTT), fibrinogen measures and platelets number (the latter is part of a classical blood cells counting at screening)
* Any inflammatory disease in the past four weeks
* Use of specific medications
* Recent major surgery (3 months)
* History of major gastro-intestinal surgery (gastric bypass, intestinal resection etc…)
* History of cancer within the past year
* Significant weight loss during the last 3 months (5% and more)
* Food allergies, especially cow milk protein allergies
* Special diets especially vegetarian, high protein or weight loss program (anamnesis)
* Smokers
* High level structured exercise 3 times a week (e.g.: fitness club, competitions…)
* Have a high alcohol consumption (more than 2 drinks/day)
* Consumption of illicit drugs anamnesis only
* Having given blood within the last month, or willing to make a blood donation until one month following the end of the study
* Subject who cannot be expected to comply with the study procedures, including consuming the test products.
* Currently participating or having participated in another clinical trial during the last month prior to the beginning of this study

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
muscle FSR determination | Within 24 hours of product intake
  Muscle protein FSR (fractional synthesis rate) will be determined using primed constant infusions of [13C6] phenylalanine for 5 hours starting around from 03:00 a.m. (see flow chart attached). Whole body protein balance will be measured throughout the night using [15N]glycine (200mg) which will be orally taken with the trial product in the evening.

SECONDARY OUTCOMES:
Activation of signaling pathways involved in skeletal muscle protein balance | Within 24 hours after product intake
  Activation of signaling pathways involved in skeletal muscle protein balance will be assessed through use of immunohistochemistry
Glucose metabolism | Within 24 hours after product intake
  Glucose metabolism will be assessed from circulating concentrations of glucose and insulin.
Plasma amino acid availability | Within 24 hours after product intake
  The quantification of Free Amino Acids in Human Plasma will be done by Amino Acid Analyser Biochrome 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic Unit, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Karagounis LG, Beaumont M, Donato-Capel L, Godin JP, Kapp AF, Draganidis D, Pinaud S, Vuichoud J, Shevlyakova M, Rade-Kukic K, Breuille D. Ingestion of a Pre-bedtime Protein Containing Beverage Prevents Overnight Induced Negative Whole Body Protein Balance in Healthy Middle-Aged Men: A Randomized Trial. Front Nutr. 2019 Nov 29;6:181. doi: 10.3389/fnut.2019.00181. eCollection 2019. PMID 31850360